CLINICAL TRIAL: NCT02355873
Title: Efficacy and Safety of Heparin-coated Surface-treated Polyacrylonitrile Membrane Hemofilter in Critical Ill CRRT Patients Continuous Renal Replacement Therapy Patients
Brief Title: Efficacy and Safety of Heparin-coated Surface-treated Polyacrylonitrile Membrane Hemofilter in Critical Ill CRRT Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Tao Su, Effect of heparin coated Surface-treated Polyacrylonitrile Membrane Hemofilter in Critical Ill CRRT Patients, Peking University First Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013QX-FZC-001
Record Dates: First submitted 2015-01-21; First posted 2015-02-04 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Critical Ill Patients; Patients Needing Continuous Renal Replacement Therapy
Keywords: heparin-coated; surface-treated polyacrylonitrile membrane hemofilter; critical ill; acute kidney injury; chronic kidney disease; continuous renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: ST100 (AN69ST) to M100 (AN69), M100 to ST100
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AN69ST (Experimental): AN69ST:Surface-treated Polyacrylonitrile Membrane Hemofilter
  Interventions: Device: AN69ST hemofilter
- AN69 (Active Comparator): AN69:original Polyacrylonitrile Membrane Hemofilter
  Interventions: Device: AN69 hemofilter

INTERVENTIONS:
Device: AN69ST hemofilter
  Arms: AN69ST
Device: AN69 hemofilter
  Arms: AN69

SUMMARY:
CRRT patients are generally critical ill patients with unstable conditions, such as low blood pressure,severe SIRS,et al. Acute kidney injury(AKI)is especially prevalent,with even two or more organ failure. CRRT serves as an important supportive therapy.Continuous anticoagulation is needed to prevent treatment interruptions due to clotting of the extracorporeal circuit. Unfractionated heparin or low molecular weight heparin both increase the risk of bleeding and heparin induced thrombocytopenia in such cases.However, the problem of CRRT without anticoagulation is the early filter clotting. An alternative method is the use of heparin coated hemofilter. The AN69 ST hemofilter, a surface-treated polyacrylonitrile membrane hemofilter, allows irreversible fixing of heparin to filter membrane, is able to reduce thrombogenic properties of the membrane. In this study, we observe the efficacy and safety of heparin-coated AN69 ST hemofilter in CRRT patients, and compare to the original AN69 membrane hemofilter.

ELIGIBILITY:
Inclusion Criteria:

* Critical ill patients who need continuous renal replacement therapy
* Continuous anticoagulation therapy is not necessarily during CRRT process

Exclusion Criteria:

* Patients needing continuous anticoagulation during each CRRT process
* Expectant survival time less than 72 hours
* Extremely unstable vital signs such as low blood pressure
* Any reasons that resulting in blood flow rate less than 150ml/min
* Pregnant women
* Patients allergic to heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The filter survival time of AN69ST and AN69 membrane hemofilter in each CRRT process | 6 months
The number of patients with early filter clotting in the scheduled CRRT using AN69ST and AN69 membrane hemofilter | 6 months
The number of patients in AN69ST and AN69 hemofilter group according to the final filter clotting grading | 6 months

SECONDARY OUTCOMES:
The number of participants with the adverse events. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renal division,department of Medcine,Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Su T, Jin Q, Liu Z. Polyethyleneimine-treated polyacrylonitrile membrane hemofilter for critically ill patients receiving anticoagulant-free prolonged intermittent renal replacement therapy: a single-center, prospective, self-controlled pilot study. BMC Nephrol. 2017 Jun 30;18(1):208. doi: 10.1186/s12882-017-0627-1. PMID 28666474